CLINICAL TRIAL: NCT02898974
Title: Medical Marijuana and Its Effects on Motor Function in People With Multiple Sclerosis: An Observational Case-control Study
Brief Title: Medical Marijuana and Its Effects on Motor Function in People With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: William R. Shaffer, M.D. (Unknown)
Responsible Party: Principal Investigator, Thorsten Rudroff, Assistant Professor, Colorado State University
Other Study IDs: 16-6685HH
Record Dates: First submitted 2016-09-06; First posted 2016-09-13 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Regular Medical Marijuana users: People with MS that are regular Medical Marijuana users
  Interventions: Behavioral: Medical Marijuana
- Non Users of Medical Marijuana: People with MS that are non users of Medical Marijuana

INTERVENTIONS:
Behavioral: Medical Marijuana — To investigate the effects of medical marijuana usage on physical function we will employ an observational case-control design
  Groups: Regular Medical Marijuana users

SUMMARY:
Medical marijuana is commonly prescribed people with Multiple Sclerosis (MS) for symptom, e.g. spasticity and pain, management. Unfortunately not much is known about its effects outside the treatment for these 2 symptoms. Several previous studies have suggested people with MS using medical marijuana have lower levels of physical disability and improved walking abilities. A major limitation of these previous studies is that the investigators used subjective measures of motor function. In this proposed observational case-control study the investigators plan to objectively measure multiple domains of motor function, such as: fatigue, strength, and walking ability. No marijuana will be brought on to campus or given to participants.

DETAILED DESCRIPTION:
To investigate the effects of medical marijuana usage on physical function the investigators will employ an observational case-control design. Cases (MS medical marijuana users) will be compared to age, sex, and disease duration matched controls (MS non-cannabis users).

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with MS,
* 30-60 years of age,
* Moderate disability (Patient Determined Disease Steps score 2-6).

Exclusion Criteria:

* Relapse with the last 60 days,
* High risk for cardiovascular disease (American College of Sports Medicine risk classification),
* Changes in disease modifying medications within the last 45 days,
* Concurrent neurological/neuromuscular disease,
* Hospitalization within the last 90 days,
* Inability to understand/sign informed consent.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults diagnosed with Multiple Sclerosis.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Rudroff, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- Department of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regular Medical Marijuana Users | Non Users of Medical Marijuana
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Medical Marijuana Users | Non Users of Medical Marijuana | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Fatigue
Description: Strength decline during fatiguing muscle contraction measured with force transducer
Time Frame: Through study completion, an average of 6 months.
Population: Twenty Two participants were enrolled in the study. Analysis was performed on sixteen people with Multiple Sclerosis, eight cannabis users and age/sex matched non-users. Matching was only possible for 16 subjects. The remaining 6 subjects were not included in the analysis.
Measure: Mean (Standard Deviation); unit: % decline
Arm/Group | Regular Medical Marijuana Users | Non Users of Medical Marijuana
Number analyzed (Participants) | 8 | 8
% decline | 21 (13) | 24 (15)

2. Primary Outcome: Muscle Strength
Description: Maximal muscle strength measured with force transducer
Time Frame: Through study completion, an average of 6 months.
Population: Twenty Two participants were enrolled in the study. Analysis was performed on sixteen people with Multiple Sclerosis, eight cannabis users and age/sex matched non-users.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Regular Medical Marijuana Users | Non Users of Medical Marijuana
Number analyzed (Participants) | 8 | 8
Newton | 28.7 (7.7) | 33.6 (10.1)

3. Primary Outcome: Postural Stability
Description: Timed up and go
Time Frame: Through study completion, an average of 6 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Regular Medical Marijuana Users | Non Users of Medical Marijuana
Number analyzed (Participants) | 8 | 8
Seconds | 9.2 (3.4) | 11.5 (13.5)

ADVERSE EVENTS:
Time Frame: Through out the study and assessed at every study visit, an average of 6 months.
Description: Twenty Two participants were enrolled in the study. Analysis was performed on sixteen people with Multiple Sclerosis, eight cannabis users and age/sex matched non-users.
Arm/Group | Regular Medical Marijuana Users | Non Users of Medical Marijuana
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT02898974/Prot_SAP_ICF_000.pdf